CLINICAL TRIAL: NCT02458170
Title: Examination of Biopsies From Healthy Knee Joints for the Use of Research Activities in Inflammatory Joint Diseases
Brief Title: Examination of Biopsies From Healthy Knee Joints
Status: Terminated | Type: Observational
Why Stopped: Shutdown of The Department of Inflammatory Diseases at Novo Nordisk.
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: N-20130026
Record Dates: First submitted 2014-09-12; First posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Abnormality in Synovial Tissue
Keywords: Rheumatoid arthritis; Synovial tissue; Joint destruction; Inflammation
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biopsies from synovial tissue.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the project is to examine what kind of molecular mechanism which causes inflammatory joint diseases. This examination is carried out by a collection and analysis of synovial tissues for patients without inflammatory joint diseases compared to the experienced equivalent biopsies from patients with inflammatory joint diseases.

DETAILED DESCRIPTION:
Arthritis is caused by autoimmune disease in the cells and pathogenesis of the tissue. This autoimmune inflammation is very often a chronic disease which causes irreversible articular damage. Rheumatoid arthritis is very often a painful and disabling disease if the treatment turns out to be ineffectual. Several of the available remedies can not treat the disease totally but only keep the patients in check.

The biological mechanisms which cause an autoimmune inflammatory articular disease have not been proved scientifically yet. Under normal conditions, the immune system adapts easily in order to protect the body against pathogenic bacteria and virus without causing damage on the body's own cells. Autoimmune inflammatory diseases displace this balance in a way so that the immune system can not distinguish between "self" and "non-self". Different kinds of cells are involved in this chronic inflammation in the joints. Majority of these cells belong to the heart of the immune response, for example T-lymphocytes, B-lymphocytes, macrophages, dendrites and granulocytes. However, other cells are also involved, for example synovial fibroblasts and endothelium.

It is very important to understand the interaction of these cells in order to develop new medicinal products for inflammatory articular diseases. The big challenge for conduction research in inflammatory articular diseases is to achieve more evidence-based knowledge of the synovial tissue from the patients and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Males and females > 18 years
* Planned surgery for patients with meniscus or reconstruction of ligament

Exclusion Criteria:

* Employment at Aalborg University Hospital
* Employment at Novo Nordisk A/S
* An unsigned statement of consent
* Current medical treatment resistant to a course of treatment, for example large doses of steroids

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohorts will be selected from primary care clinic.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Adverse events as a measure of metabolism in normal tissue and inflammatory tissue. | 7 years
  Compare the normal metabolism in non-inflammatory tissue with biopsies of inflammatory diseases.

SECONDARY OUTCOMES:
Detect new objects for developing drugs. | 7 years
  Determine potential objects for medical intervention and development of drugs which affect the molecular mechanisms in relation to an inflammatory condition versus a normal metabolic condition.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, M.D., Study Chair — Northern Orthopaedic Division, Aalborg University Hospital
Locations (1):
- Northern Orthopaedic Division, Aalborg University Hospital, Aalborg, Denmark